CLINICAL TRIAL: NCT02552953
Title: A Phase I Pharmacologic Study of CYC065, a Cyclin Dependent Kinase Inhibitor, in Patients With Advanced Cancers
Brief Title: A Pharmacologic Study of CYC065, a Cyclin Dependent Kinase Inhibitor, in Patients With Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cyclacel Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYC065-01
Record Dates: First submitted 2015-09-11; First posted 2015-09-17 (Estimated); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — CYC065

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CYC065 - 4 hour infusion (Part 1 completed) (Experimental): CYC065 will be administered by 4 -hour infusion every 3 weeks.
  Interventions: Drug: CYC065
- CYC065 - 1 hour infusion (Part 2 - ongoing) (Experimental): CYC065 will be administered by 1 - hour infusion on Days 1, 2, 8, and 9 every 3 weeks
  Interventions: Drug: CYC065
- CYC065 - Oral (Part 3 - ongoing) (Experimental): CYC065 will be administered orally on Days 1, 2, 8 and 9 every 3 weeks
  Interventions: Drug: CYC065

INTERVENTIONS:
Drug: CYC065

SUMMARY:
This is an open-label, single arm, dose escalation study in patients with advanced cancers.

DETAILED DESCRIPTION:
This is an open-label, single arm, dose escalation study in patients with advanced cancers. Treatment will be administered on an outpatient basis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumors or lymphomas that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* 18 years or older
* ECOG performance status 0-1
* Life expectancy ≥ 3 months
* Evaluable disease
* Adequate organ functions
* 4 weeks from prior chemotherapy ( 6 weeks for mitomycin C and nitrosourea) , immunotherapy, investigational anti-cancer therapy, radiation therapy; and have recovered from prior toxicities
* At least 4 weeks from major surgery
* Agree to practice effective contraception
* Agree to follow protocol required evaluations
* Ability to understand and willingness to sign the informed consent form

Exclusion Criteria:

* Previously untreated CNS metastasis or progressive CNS metastasis
* Currently receiving radiotherapy, biological therapy, or any other investigational agents
* Uncontrolled intercurrent illness
* Pregnant or lactating women
* Known to be HIV-positive
* Known active hepatitis B and/or hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Number of patients who experience dose-limiting toxicities | cycle 1(each cycle is 21 -28 days)

SECONDARY OUTCOMES:
Plasma concentrations | cycle 1(each cycle is 21 -28 days)
Half-life of CYC065 | cycle 1(each cycle is 21 -28 days)
changes in certain protein levels in peripheral white blood cells by western blots | cycle 1(each cycle is 21 -28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Shapiro, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States